CLINICAL TRIAL: NCT03970759
Title: A Review of Meta-Analyses on Bioavailable Stannous Fluoride Dentifrices: Effects on Gingival Health
Brief Title: Meta-analysis of Stannous Fluoride and the Effects on Gingival Health
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019SnF2GIAnalysis
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stannous Fluoride Dentifrice: Twice daily brushing
  Interventions: Drug: Stannous Fluoride Dentifrice
- Positive Control Dentifrice: Twice daily brushing
  Interventions: Drug: Positive control dentifrice
- Negative Control Dentifrice: Twice daily brushing
  Interventions: Drug: Negative control dentifrice

INTERVENTIONS:
Drug: Stannous Fluoride Dentifrice — Experimental stannous fluoride (0.454%) dentifrice
  Groups: Stannous Fluoride Dentifrice
Drug: Positive control dentifrice — Positive control dentifrice containing (0.3%) triclosan.
  Groups: Positive Control Dentifrice
Drug: Negative control dentifrice — Negative control dentifrice containing either sodium fluoride (0.243%) or sodium monofluorophosphate (0.76%)
  Groups: Negative Control Dentifrice

SUMMARY:
The aim of this 18 study analysis was to compare the effect of bioavailable stannous fluoride (SnF2) dentifrices when used up to 3 months on gingivitis relative to a positive or negative control dentifrice.

ELIGIBILITY:
Subjects were excluded from this study for the following reasons;

* pregnancy,
* rampant caries,
* severe periodontitis,
* at discretionary of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females with mild-moderate gingivitis.
Sampling Method: Probability Sample
Enrollment: 2890 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Bleeding Sites | Up to 12 Weeks
  Change from baseline as measured on number of bleeding sites (gingival bleeding index or Loe Silness index).

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple P&G Investigation Clinical Sites, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Biesbrock A, He T, DiGennaro J, Zou Y, Ramsey D, Garcia-Godoy F. The effects of bioavailable gluconate chelated stannous fluoride dentifrice on gingival bleeding: Meta-analysis of eighteen randomized controlled trials. J Clin Periodontol. 2019 Dec;46(12):1205-1216. doi: 10.1111/jcpe.13203. PMID 31562774